CLINICAL TRIAL: NCT07120074
Title: The Effects Of Dual-Task Exercises On Balance And Cognitive Function In Individuals With Different Physical Performance Levels
Brief Title: Dual-Task Exercise Effects on Balance and Cognition by Physical Performance Level
Acronym: Dual Task
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Tulin Unal, Physiotherapist, Bahçeşehir University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: -78097791-020-4138; Bahcesehir University (Other: Bahcesehir University)
Record Dates: First submitted 2025-07-20; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Dual Task; Physical Activity Levels
Keywords: dual task; denge
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants aged between 20 and 50 years were divided into two groups based on their physical performance levels. Both groups performed dual-task exercises.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Highly active dual-task exercise group (Active Comparator): Dual-task exercises involve the simultaneous performance of a motor task (e.g., walking, balancing, carrying an object) and a cognitive task (e.g., counting, word recall, attention tasks). These exercises simulate real-life situations that require multitasking and aim to improve motor-cognitive integration. They have been shown to be effective in enhancing balance, gait, and cognitive functions, particularly in older adults, individuals with neurological disorders, and those at risk of falling.Based on the International Physical Activity Questionnaire - Short Form (IPAQ-SF) scores, participants were categorized into two groups: highly active and less active. Both groups underwent the same dual-task exercise protocol.
  Interventions: Other: Exercise
- Low-activity dual-task exercise group (Active Comparator): Dual-task exercises involve the simultaneous performance of a motor task (e.g., walking, balancing, carrying an object) and a cognitive task (e.g., counting, word recall, attention tasks). These exercises simulate real-life situations that require multitasking and aim to improve motor-cognitive integration. They have been shown to be effective in enhancing balance, gait, and cognitive functions, particularly in older adults, individuals with neurological disorders, and those at risk of falling. Based on the International Physical Activity Questionnaire - Short Form (IPAQ-SF) scores, participants were categorized into two groups: highly active and less active. Both groups underwent the same dual-task exercise protocol.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — A low-activity exercise group, and highly active dual-task exercise group determined based on physical performance level, was subjected to 6 weeks of dual-task exercises aimed at improving balance and cognitive function. Dual-task refers to performing two different tasks simultaneously. In the first week, tasks included generating 3- and 4-letter words while standing in a tandem position, reciting the months and seasons in order while shifting weight forward and backward on a balance board, and performing addition and subtraction tasks while walking. The difficulty level of the tasks was increased each week.

SUMMARY:
This study aims to investigate the effects of dual-task exercises on balance and cognitive function in individuals with varying levels of physical performance. Dual-task training, which involves performing cognitive and motor activities simultaneously, has been shown to improve functional mobility, especially in older adults and patients with neurological conditions. However, limited data exist on how these effects differ among individuals with different physical capacities. The findings of this study will contribute to understanding the therapeutic value of dual-task exercises in promoting both physical and cognitive health.

DETAILED DESCRIPTION:
Physical activity is a fundamental element of a healthy lifestyle, playing a critical role in improving overall health and enhancing long-term quality of life. Defined as any bodily movement produced by skeletal muscles that results in energy expenditure, physical activity encompasses a broad range of behaviors, including household chores, leisure-time sports, school physical education, and structured exercise. Exercise, a subset of physical activity, refers to planned, repetitive, and purposeful movement aimed at improving physical fitness. The frequency, intensity, and duration of activity are key factors in its classification and effectiveness. Physical activities can also be categorized by context-such as those occurring during work, sleep, or leisure time-with leisure-time activities further divided into exercise, sports, domestic chores, and other tasks.

Daily life often requires performing multiple tasks at the same time, placing simultaneous demands on both motor and cognitive functions. Dual-task training, which evaluates the ability to perform cognitive and motor activities concurrently, is gaining increasing attention. In recent years, shifts in occupational and lifestyle demands-driven by technological advancement-have led to increased reliance on cognitive skills, underscoring the importance of dual-task capacity in modern life.

Research has shown that performing simultaneous tasks can challenge attentional resources, particularly when cognitive and motor demands are high. This can lead to decreased performance, a phenomenon referred to as dual-task interference. Such interference is influenced by multiple factors, including task difficulty, attentional demands, task prioritization, and individual characteristics like age, fear of falling, and cognitive or motor abilities.

Balance control depends on the integration of visual, vestibular, and somatosensory inputs, alongside neuromuscular feedback. It is fundamental to the performance of voluntary motor actions and is affected by environmental context and task specificity.

The literature demonstrates that dual-task training has been effective in older adults, improving functions such as gait, balance, and reducing fall risk. Studies involving patients with neurological conditions (e.g., Parkinson's disease) also highlight improvements in motor and cognitive performance following dual-task interventions. These gains have been associated with greater autonomy in activities of daily living.

Despite these promising outcomes, few studies have examined the effects of dual-task training across populations with different physical performance levels. Our study aims to address this gap by evaluating how individuals with varying physical capacities respond to dual-task exercise programs in terms of balance and cognitive function. The overarching goal is to contribute to evidence supporting the integration of dual-task interventions into broader health promotion and rehabilitation strategies targeting both physical and mental well-being.

ELIGIBILITY:
Inclusion Criteria:

Aged between 20 and 50 years Adequate cognitive function to understand instructions and participate in the study Willingness and ability to participate regularly in the exercise program Ability to comprehend and follow the study procedures

Exclusion Criteria:

Diagnosed with rheumatoid arthritis Diagnosed with systemic lupus erythematosus (SLE) Diagnosed with Parkinson's disease Diagnosed with multiple sclerosis History of stroke Diagnosed with Alzheimer's disease or other dementias Diagnosed with scoliosis causing physical limitation History of lower limb fractures Presence of foot or ankle tendonitis Diagnosed with color blindness or legal blindness History of major surgery (e.g., orthopedic, spinal, abdominal) within the past 6 months Irregular attendance or non-compliance with the exercise protocol

Ages: 20 Months to 50 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2025-08-03 (Estimated); Primary Completion 2025-10-04 (Estimated); Study Completion 2025-11-18 (Estimated)

PRIMARY OUTCOMES:
Single-Leg Stance Test | At baseline and after 6 weeks
  First, the participant will be asked which foot they prefer to stand on or which foot makes them feel more stable. Then, they will be instructed to distribute their weight evenly on both feet and, while maintaining this position, lift one foot off the ground. The timer will start as soon as the participant lifts their foot. The timer will be stopped if any signs of balance disturbance occur, such as the lifted foot making contact with the ground, the standing foot jumping, or the participant needing to support themselves in order to maintain balance. The longer an individual is able to maintain a single-leg stance, the better their static balance is considered to be.
Y Balance Test | At baseline and after 6 weeks exercise program
  The Y-Balance Test (YBT) is a widely used, valid, and reliable tool for assessing dynamic balance. In this test, the participant stands on one leg and reaches in specific directions (anterior, posteromedial, and posterolateral) with the opposite leg. In this study, only the anterior reach direction was assessed.
  Participants performed three practice trials for familiarization, followed by three recorded trials. During the test, the participant stood barefoot on a flat surface, maintaining balance on one leg. With the contralateral leg, they reached forward as far as possible and returned to the starting position without losing balance. The distance was measured from the tip of the big toe of the stance foot to the point where the toes of the reaching foot touched the ground. The longest distance achieved among the trials was used for statistical analysis.
  Greater reach distances were interpreted as better dynamic balance performance.
Stroop Test | At baseline and after 6 weeks exercise program
  The aim of the Stroop test is to evaluate the person's speed of processing information, especially simple and complex attention, inhibition ability, ability to be resistant to interference. The test to be used in our study includes 3 steps: In the first step, the person is asked to say the colours of the boxes in the form, in the second step to read the words in the form quickly, and in the last step to say the colours of the words. The time taken to complete each step is noted. The time difference between steps 2 and 3, the error made and the self-correction scores are recorded.

SECONDARY OUTCOMES:
Health-Related Quality of Life assessed by the SF-36 Questionnaire | At baseline and after 6 weeks exercise program
  The SF-36 questionnaire is a quality of life questionnaire that includes 36 questions divided into 8 different categories (physical functioning, limitations due to physical condition, physical pain, perceived health, vitality, social functioning or well-being, limitations due to mental condition, mental health). These 8 dimensions are used to calculate two scores on the quality of life of individuals: the physical composite score and the mental composite score. The higher the score, the greater the capacity. It is self-administered and takes less than 10 minutes. Higher scores indicate better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: tulin unal, Principal Investigator — bağlantısız
Locations (1):
- Bahcesehir University, Istanbul, MALTEPE, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Anonymized demographic information of participants (e.g., age, gender, educational status) Balance assessment scores before and after dual-task exercises Cognitive function assessment results (Stroop test) Quality of life evaluation results (SF-36)
Supporting Information: Study Protocol, SAP